CLINICAL TRIAL: NCT04828941
Title: A 26-week Randomized Clinical Trial of an Electronic Headache Diary in Migraine Patients
Brief Title: My Healthy Diary - An Electronic Diary for Remote Migraine Monitoring
Acronym: E-Migra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Matosinhos, EPE (Other)
Responsible Party: Principal Investigator, Axel Ferreira, MD, PhDs, Unidade Local de Saúde de Matosinhos, EPE
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 96/CE/JAS
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Episodic Migraine; Migraine Disorders
Keywords: Migraine Disorders; mHealth; Mobile Applications; Health Diaries
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Each patient will use the electronic headache diary and the paper diary for a period of 13 weeks, the order of their use will be determined by randomisation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Headache Diary (Experimental): The electronic headache diary registers: total number of days with headache per month, number of days with migraine per month, number of days with tension headache per month, number of days taking SOS medication per month, number of days with incapacity for work per month, number of days in which patient goes to the emergency department.
  Interventions: Device: Electronic Headache Diary
- Paper Diary (Active Comparator): The paper headache diary registers: total number of days with headache per month, number of days with migraine per month, number of days with tension headache per month, number of days taking SOS medication per month, number of days with incapacity for work per month, number of days in which patient goes to the emergency department.
  Interventions: Device: Paper Diary

INTERVENTIONS:
Device: Electronic Headache Diary — The electronic headache diary is an app-based diary that permits the registration of headaches, their acute treatment and their associated work incapacity. It also permits real-time monitoring of these data.
  Arms: Electronic Headache Diary
Device: Paper Diary — The paper diary permits the registration of the same variables as the electronic diary in paper format.
  Arms: Paper Diary

SUMMARY:
This study aims to evaluate the usefulness of an app-based headache diary in episodic migraine patients. For this the investigators will conduct a randomized clinical trial with a crossover design, using the app-based diary and a traditional paper-based headache diary. The patients will use each diary for 13 weeks. The investigators will evaluate diary adhesion after each 13-week period, and also evaluate headache burden and prophylactic medication compliance at the beginning, at the crossover point, and at the end of the study, and acute headache medication use through diary records. The investigators will also evaluate user preference through a questionnaire at the end of the study.

DETAILED DESCRIPTION:
Headache is one of the main reasons for seeking primary health care and an important cause of absenteeism at work and decreased quality of life in the population, being the major neurological cause of disability in young adults and middle-aged adults. Although the subjectivity of the complaints and the great intra and inter-individual variability of clinical presentations hinder its epidemiological study, it is estimated that the overall prevalence of headache throughout life is 66% (46-78% in tension-type headache; 14-16% for migraine and 0.1-0.3% for cluster headache). Migraine, in particular, is a primary headache with an estimated prevalence of 11 to 14% in adult women and 4 to 9% in adult men. In addition, it is assumed that up to 20% of absences from work can be attributed to headaches, with the inherent socio-economic impacts.

Headache is a very frequent complaint in the primary care setting. However, the differential diagnosis can be complicated at this level. Primary headache diagnosis is made almost exclusively through clinical history taking, for this purpose clinicians use the criteria in the International Classification of Headache Disorders, currently on its 3rd version. However, its application is often challenging and time-consuming, especially in a primary care setting, where physicians are very limited on time. Nonetheless, a correct diagnosis is essential, as treatment varies among the primary headaches and also within the same headache type according to its frequency.

The episodic nature of headaches increases the risk of memory bias towards more severe or more recent crises. To avoid this, patients nowadays use a paper calendar. This calendar makes it possible to monitor, more reliably, the response to therapy and to identify the need for any adjustments.

However, the paper calendar has many limitations, such as the possibility of filling in immediately before consultations instead of non-biased daily records. In addition, the paper or card used can be lost, is more easily forgotten, and cannot be consulted remotely by the attending physician. In the current digital landscape, we have seen a transition in registration methods for semi-automated electronic platforms, considered more practical and appealing to users. However, most in-app headache diaries are not validated and are mainly written in English.

Having these ideas in mind the investigators decided to develop an app-based electronic headache diary that would not only permit a better adhesion to follow-up but also remote monitoring of headache patients. To study the applicability and the usefulness of this idea the investigators designed a randomized clinical trial with a crossover design where episodic migraine patients would be randomized to the use of the app or of a paper headache diary. Each patient would use the app and the paper diary for a period of 13 weeks.

In the paper and electronic diary patients will record headache days, headache type (migraine or tension-type headache), headache intensity with a scale from 0 to 10, intake of acute headache medication, missing work days due to headache, and recurrence to the emergency department due to headache.

The investigators will also measure headache burden with the portuguese versions of HIT-6, MSQ v2.1 and MiDAS scales and quality of life with the WHOQOL-BREF at the beginning, at the crossover point, and at the end of the study. Also, the study will evaluate prophylactic medication compliance at the beginning, at the crossover point, and at the end of the study through a questionnaire. User preference will be measured through a questionnaire, using a Likert type scale, at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with episodic migraine, diagnosed for more than 6 months.
* Patients with at least 4 headache days per month and a maximum of 15 headache days per month.

Exclusion Criteria:

* Patients with major psychiatric illness.
* Patients participating in another clinical trial.
* Patients who do not meet diagnostic criteria for episodic migraine according to ICHD-3.
* Illiterate patients or those who are unable to fill the records independently.
* Patients with a previous history of filling in a headache calendar, in the 3 months prior to randomization.
* Patients who do not use a cell phone with Android OS.
* Patients who cannot read or write in Portuguese.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-28 (Estimated); Primary Completion 2021-10-02 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Diary compliance | 6 months
  To assess whether the compliance of migraine patients to the use of an electronic headache diary is superior to adherence to the paper diary. The quantification of adherence will be made in: 1.1.) % Of days per month of headache registration; and 1.2.) % of patients who abandon calendar registration at 13 weeks.

SECONDARY OUTCOMES:
Patient Preference | 6 months
  Preference of the patient for one of the diaries measured through a questionnaire.
Quality of Life (HIT-6) | 6 months
  Comparison of the quality of life using data from HIT-6 evaluated at the baseline, after using the electronic diary and after using the paper diary.
Quality of Life (MSQ v2.1) | 6 months
  Comparison of the quality of life using data from MSQ v2.1 evaluated at the baseline, after using the electronic diary and after using the paper diary.
Quality of Life (WHOQOL-BREF) | 6 months
  Comparison of the quality of life using data from WHOQOL-BREF evaluated at the baseline, after using the electronic diary and after using the paper diary.
Incapacity Days | 6 months
  Comparison of the number of incapacity days using data from the diaries and from MiDAS evaluated at the baseline, after using the electronic diary and after using the paper diary.
Subjective Evaluation of the Number of Headache Days | 6 months
  Comparison of the patient's subjective evaluation of the number of headache days using data from questionnaires evaluated at the baseline, after using the electronic diary and after using the paper diary.
Number of Acute Headache Medication Use Days | 6 months
  Comparison of the number of acute headache medication use days using data from the diaries and questionnaires filled at the baseline, after using the electronic diary and after using the paper diary.
Prophylactic Medication Compliance | 6 months
  Comparison of the number of days of prophylactic medication noncompliance evaluated by questionnaire at the baseline, after using the electronic diary and after using the paper diary.
Emergency Department Visits | 6 months
  Comparison of the number of emergency department visits evaluated by data collected from the diaries and a questionnaire filled at the baseline, after using the electronic diary and after using the paper diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pedro Hispano, Unidade Local de Saúde de Matosinhos, Matosinhos Municipality, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becker WJ, Findlay T, Moga C, Scott NA, Harstall C, Taenzer P. Guideline for primary care management of headache in adults. Can Fam Physician. 2015 Aug;61(8):670-9. PMID 26273080
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Nappi G, Jensen R, Nappi RE, Sances G, Torelli P, Olesen J. Diaries and calendars for migraine. A review. Cephalalgia. 2006 Aug;26(8):905-16. doi: 10.1111/j.1468-2982.2006.01155.x. PMID 16886925
- [Background] Baos V, Ester F, Castellanos A, Nocea G, Caloto MT, Gerth WC; I-Max Study Group. Use of a structured migraine diary improves patient and physician communication about migraine disability and treatment outcomes. Int J Clin Pract. 2005 Mar;59(3):281-6. doi: 10.1111/j.1742-1241.2005.00469.x. PMID 15857323
- [Background] Allena M, Cuzzoni MG, Tassorelli C, Nappi G, Antonaci F. An electronic diary on a palm device for headache monitoring: a preliminary experience. J Headache Pain. 2012 Oct;13(7):537-41. doi: 10.1007/s10194-012-0473-2. Epub 2012 Jul 28. PMID 22842873
- [Background] Hundert AS, Huguet A, McGrath PJ, Stinson JN, Wheaton M. Commercially available mobile phone headache diary apps: a systematic review. JMIR Mhealth Uhealth. 2014 Aug 19;2(3):e36. doi: 10.2196/mhealth.3452. PMID 25138438
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Martin BC, Pathak DS, Sharfman MI, Adelman JU, Taylor F, Kwong WJ, Jhingran P. Validity and reliability of the migraine-specific quality of life questionnaire (MSQ Version 2.1). Headache. 2000 Mar;40(3):204-15. doi: 10.1046/j.1526-4610.2000.00030.x. PMID 10759923
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902